CLINICAL TRIAL: NCT05413811
Title: Acceptability and Feasibility of Combination Treatment for Cervical Precancer Among South African Women Living With HIV
Acronym: ACT2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IGHID12046; 1R01CA250850-01 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer; CIN2; CIN3; Human Immunodeficiency Virus; Human Papillomavirus
Keywords: 5-fluorouracil cream; Loop electrosurgical excision
MeSH Terms: conditions — Uterine Cervical Neoplasms; Acquired Immunodeficiency Syndrome | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5 Fluorouracil Cream (Experimental): The participants will receive 8 doses of intravaginal 5 Fluorouracil Cream.
  Interventions: Drug: 5 Fluorouracil (5 FU) Cream
- Placebo Cream (Placebo Comparator): The participants will receive 8 doses of intravaginal placebo cream.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5 Fluorouracil (5 FU) Cream — Intravaginal topical chemotherapy, 5-fluorouracil cream
  Other Names: Fluoroplex; Efudex; Carac
  Arms: 5 Fluorouracil Cream
Drug: Placebo — Intravaginal topical placebo cream
  Arms: Placebo Cream

SUMMARY:
The purpose of this study is to explore whether an anti-cancer medication (5-fluorouracil cream) placed in the vagina after a surgical excision procedure is an acceptable and useful form of treatment for cervical precancer among the woman with HIV infection.

DETAILED DESCRIPTION:
There are currently no medical therapies recommended to promote the clearance of humanpapilloma virus (HPV) infection, regression of cervical dysplasia, or treatment of cervical intraepithelial neoplasia (CIN). Human immunodeficiency virus (HIV) -infected women are at higher risk of HPV infection, with rates as high as 45% - 90%. Despite being preventable, cytologic abnormalities, cervical precancer (high-grade cervical intraepithelial neoplasia [CIN2/3]), and invasive cervical cancer also occur more frequently in HIV infected women.

This study is testing whether topical 5-fluorouracil (5FU) can be used as a patient-controlled adjuvant treatment for cervical precancer (CIN2/3) to be self-administered after surgical excision to reduce the risk of persistent/recurrent CIN2/3 and progression to cervical cancer among HIV-infected women.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection
* On antiretroviral therapy (ART), for at least 90 days prior to enrollment
* Cervical biopsy demonstrating CIN2/3 within the preceding 120 days.

Exclusion Criteria:

* pregnancy,
* breastfeeding,
* intend to become pregnant within 180 days of enrollment
* have an active sexually transmitted infection (women may participate once treated)
* have a surgically absent cervix
* have a history of anogenital (cervical, vaginal, vulvar, or anal) cancer or a biopsy suspicious for cervical cancer
* have a medical comorbidity that would interfere with study participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The target population is HIV-infected women only.
Enrollment: 180 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-08-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
The number of subjects adhered to and retained in the study | Up to 24 weeks
  The feasibility of the combination of surgical excision followed by adjuvant 5FU for the treatment of CIN2/3 among HIV-infected women will be evaluated using the number of subjects adhered to and retained in the study.
The number of participants who found the intervention acceptable | week 10 to week 24
  The acceptability of the combination of surgical excision followed by adjuvant 5FU for the treatment of CIN2/3 among HIV-infected women will be assessed through a participant questionnaire administered at midline and end of the study.

SECONDARY OUTCOMES:
The proportion of participants with CIN2 or CIN 3 that regressed to CIN1 | 24 weeks
  Efficacy of combination treatment for CIN2/3 will be assessed as the number of subjects with CIN2 or CIN3 regressed to CIN1 or normal histology.
The percentage of participants who demonstrate clearance of high-risk HPV | 24 weeks
  Efficacy of combination treatment for HPV will be assessed as the percentage of women in each study arm who demonstrate clearance of high-risk HPV between baseline and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Chibwesha, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Clinical HIV Research Unit Temba Lethu Wing Helen Joseph Hospital, Westdene, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No
The rights and privacy of individuals who participate in research will be protected at all times. Thus, data intended for broader use will be stripped of identifiers that would permit linkages to individual research participants or variables that could lead to deductive disclosure of the identity of individual subjects. Research data that documents, supports and validates research findings will be made available after the main findings from the final research dataset have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers. All data sharing will abide by rules and/or policies defined by the sponsor, relevant IRBs, U.S. local, state, and federal laws and regulations, as well as South African laws and regulations.

REFERENCES:
- [Derived] Chibwesha CJ, Mollan KR, Teodoro NS, Keys JR, Liu C, Mulongo M, Gumede S, Pasipamire T, Faesen M, Rahangdale L. ACT 2 Clinical Trial Design: Acceptability and Feasibility of Combination Treatment for Cervical Precancer Among South African Women Living with HIV. medRxiv [Preprint]. 2025 Aug 14:2025.08.12.25333540. doi: 10.1101/2025.08.12.25333540. PMID 40832398
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials